CLINICAL TRIAL: NCT05469438
Title: IMAS Optimization and Applicability in Acute and Subacute Stroke.
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Ciro Ramos Estebanez, MD., Ph.D., Clinical Professor, Case Western Reserve University
Other Study IDs: STUDY20190922
Record Dates: First submitted 2022-03-16; First posted 2022-07-21 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acute Stroke
Keywords: Stroke; Rehabilitation; Motor Recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator will investigate our Integrated sensor-based Motion Analysis Suite (IMAS) to objectively and quantitatively measure acute stroke patient motor status.

DETAILED DESCRIPTION:
The investigator will evaluate the feasibility of our IMAS to assess 30 stroke subjects in 5 sessions (the first 4 proximal to stroke onset and the last session ~6-8 weeks post stroke). The investigator will test IMAS in 30 acute stroke subjects; and extract quantitative movement kinematic/kinetic metrics descriptive of subjects' motor behavior (e.g., arm movement speed, smoothness). Subjects will undergo a series of upper limb focused assessments including Fugl Meyer, Barthel Index, and Orpington Prognostic Scale assessments. The investigator will also collect demographics, and stroke clinical information such as imaging data.

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent to participate in the study.
2. Age 18 to 85 years old.
3. Clinical presentation and neuroimaging (CTA-CTP/ MRI-MRA) consistent with the diagnosis of Acute Ischemic or Hemorrhagic Stroke.
4. Preserved mental status (Glasgow coma score >12: E(4), V(5), M (4-6)).
5. Presence of upper limb weakness per the NIHSS (1-2 points in the arm) and ability to perform testing (i.e., NIHSS motor score 1-2 at elbow, wrist, and finger flexion-extension) within 30 days from stroke. (Note that individuals with a prior ischemic or hemorrhagic stroke with available information pertaining superior extremity baseline strength after their previous stroke would qualify).
6. Presence of upper limb weakness per the NIHSS (2 points in the arm) and ability to perform testing (i.e., NIHSS motor score 2 at elbow, wrist, and finger flexion-extension) in subacute stroke. (Note that individuals with a prior ischemic or hemorrhagic stroke with available information pertaining superior extremity baseline strength after their previous stroke would qualify).
7. Baseline Modified Rankin score <4.

Exclusion Criteria

1. History of dementia per relative/ medical records.
2. Presence of receptive aphasia at baseline or after the current acute stroke.
3. Need for rapid clinical response due to conditions such as psychosis, or suicidality.
4. Unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, pulmonary issues, or chronic obstructive pulmonary disease);
5. Amputated limbs.
6. Absence of weakness as per the NIHSS (0 points = no drift for motor arm and leg items) or severe motor impairment NIHSS 4 points for motor arm).
7. Stroke mimics (e.g., infections, medication effects from sedatives, electrolyte imbalances, etc.).
8. Stroke worsening between assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presence of upper limb weakness per the NIHSS (1-2 points in the arm) and ability to perform testing (i.e. NIHSS motor score 1-2 at elbow, wrist, and finger flexion extension)..
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ciro Ramos Estebanez, MD., Ph.D., MBA, FNCS., Chicago, Illinois
  - UH, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 consented, 8 did not meet eligibility, and 30 were enrolled and started.
Groups:
- Single Arm: Single Arm Stroke Study
Period: Overall Study
Arm/Group | Single Arm
Started (Patients that underwent at least 1 IMAS testing session) | 30
Completed (Patients that underwent at least 1 IMAS testing session) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30 Acute or Sub Acute Stroke Patients
Groups:
- Single Arm Stroke Study: 30 Acute or Sub Acute Stroke Patients
Arm/Group | Single Arm Stroke Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.96 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Fugl-Meyer [Mean (Standard Deviation); unit: units on a scale] — Upper Limb Fugl-Meyer Score (range: 0-54 ) built from a total of:
  * Volitional movement within synergies: 0-18 points
  * Volitional movement mixing synergies: 0-6 points
  * Volitional movement with little/no synergy: 0-6 points
  * Hand: 0 -14 points
  * Wrist: 0 - 10 points Higher values represent a better outcome
  units on a scale | 45.6 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: Coefficient of Determination (R²) for Predicting Fugl-Meyer Upper Extremity Score Recovery Post-stroke.
Description: The coefficient of determination (R²) quantifies how well the predictive model explains variance in Fugl-Meyer Upper Extremity recovery scores. This unitless measure ranges from -∞ to 1, with higher values indicating better model fit (i.e. better prediction).
  Additional Detail: A sensor suite assessed movement kinematics (e.g., time, position, velocity), and software predicted recovery from baseline characteristics. We report R² for the best-performing model predicting end-of-study FM score from day-one FM score, using leave-one-out cross-validation (~24 degrees of freedom). Models with fewer degrees of freedom may yield lower R² due to overfitting control.
Time Frame: 6 - 8 weeks post acute stroke onset
Population: Patients with stroke
Measure: Number; unit: Coefficient of determination (Unitless)
Groups:
- Single Arm: Single Arm- no intervention
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Coefficient of determination (Unitless) | 0.9
Statistical Analysis 1: Comparison: Single Arm; Test type: Other — We assessed prediction accuracy of our system using the R^2 from leave-one-out cross-validation of predicted Fugl-Meyer scores, which were obtained from models predicting recovery based on baseline data; We assessed prediction accuracy of our system using the R^2 from leave-one-out cross-validation of predicted Fugl-Meyer scores, which were obtained from models predicting recovery based on baseline data

ADVERSE EVENTS:
Time Frame: Occurrence of adverse events was assessed at all visits through study completion, an average of 8 weeks.
Description: There were no adverse events.
Arm/Group | Single Arm Stroke Study
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a generic non-disclosure agreement about the IMAS technology.

DOCUMENTS (2):
  • Study Protocol (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05469438/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT05469438/SAP_001.pdf